CLINICAL TRIAL: NCT03672513
Title: Short-term Supplementation, Bone Turnover and Antioxidant Status in Postmenopausal Stage: A Placebo Controlled Study.
Brief Title: Short-term Supplementation, Bone Turnover and Antioxidant Status in Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Elena Planells del Pozo, University Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FA COST Action TD1304
Record Dates: First submitted 2018-09-08; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Menopause; Nutritional Intervention; Bone Diseases
Keywords: Menopuase; Zinc; Magnesium; Antioxidant; Bone loss; Nutritional intervention
MeSH Terms: conditions — Bone Diseases; Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Supplemented Group (Placebo Comparator): Placebo control
  Interventions: Dietary Supplement: Placebo Comparator
- Magnesium Supplemented Group (Experimental): Magnesium Group
  Interventions: Dietary Supplement: Magnesium supplement
- Zinc Supplemented Group (Experimental): Zinc Group
  Interventions: Dietary Supplement: Zinc Supplement

INTERVENTIONS:
Dietary Supplement: Placebo Comparator — Oral administration of 1 daily capsule containing lactose
  Arms: Placebo Supplemented Group
Dietary Supplement: Zinc Supplement — Oral administration of 1 daily capsule containing 50 mg/day of Zn
  Arms: Zinc Supplemented Group
Dietary Supplement: Magnesium supplement — Oral administration of 1 daily capsule containing 500 mg/day of Magnesium
  Arms: Magnesium Supplemented Group

SUMMARY:
This is a 8-week, double-blinded, placebo-controlled, randomized intervention trial to investigate the effects of Mg and Zn supplementation on antioxidant status and bone hormonal parameters. Participants were randomly assigned to one of three treatment groups: Placebo group (PbG: 25 women); Magnesium Group - 500 mg/day of Mg (MgG: 27 women); Zinc Group - 50 mg/day of Zn (ZnG: 26 women).

DETAILED DESCRIPTION:
Seventy-eight healthy postmenopausal volunteers aged between 44 and 76 were recruited once had been informed about the protocol. This is a 8-week, double-blinded, placebo-controlled, randomized intervention trial to investigate the effects of Mg and Zn supplementation on antioxidant status and bone hormonal parameters. Participants were randomly assigned to one of three treatment groups: Placebo group (PbG: 25 women); Magnesium Group - 500 mg/day of Mg (MgG: 27 women); Zinc Group - 50 mg/day of Zn (ZnG: 26 women).

ELIGIBILITY:
Inclusion Criteria:

* to present postmenopausal status (with at least 12 months of amenorrhea)
* to present low status in Mg and/or Zn obtained in a previous biochemical assessment
* not present any pathology that could affect their nutritional status
* not to be subjected to hormone replacement therapy (HRT)
* not to demonstrate lactose intolerance

Exclusion criteria

* acute or terminal illness
* unwillingness to either complete the study requirements or to be randomised into control or experimental group
* to be smoker
* to be on a medication regimen

Ages: 44 Years to 76 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female, Adult
Enrollment: 78 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-09-08 (Actual)

PRIMARY OUTCOMES:
Antioxidant status | 2 months
  Total antioxidant capacity (TAC) determination in plasma samples was carried out evaluating the reduction power of Cu2+ from the action of antioxidants present in samples (TAC kit, Jaica, Shizuoka, Japan). Values were expressed in umol/L.
Oxidative stress | 2 months
  Glutathione peroxidase (GPx) in mU/mL and Superoxide dismutase (SOD) in U/mL. GPx activity was determined by using the Bioxytech GPx-340™ kit (OxisResearch™), an indirect colorimetric assay of the activity of c-GPx [28]. SOD activity was determined by using the Randox Ransod kit (RANDOX Laboratories Ltd., United Kingdom).

SECONDARY OUTCOMES:
Anthropometric assessment - Height | 2 months
  Values were expressed in centimeters.
Anthropometric assessment - Waist circumference | 2 months
  Values were expressed in centimeters.
Anthropometric assessment - Body composition by bioelectrical impedance | 2 months
  Body composition assessment was taken by multifrequency bioelectrical impedance (Tanita MC-980 Body Composition Analyzer MA Multifrequency Segmental, Barcelona, Spain). The analyzer complies with the applicable European standards (93/42EEC, 90/384EEC) for use in the medical industry. Participants were informed in advance of the required conditions prior to the measurement: no alcohol less than 24 hours before the measurement, no vigorous exercise less than 12 hours prior to the measurement, no food or drink less than 3 hours prior to the measurement, and no urination immediately before the measurement. All measurements were taken simultaneously during the morning in fasting conditions. The following measurements were taken: weight, body mass index (calculated as weight/height^2 and expressed kg/m2) and fat mass (expressed in kilograms and as the percentage of body fat), fat free mass (expressed in kilograms and as the percentage of fat free mass), muscle mass (expressed in kilograms).
Intake assessment | 2 months
  Dietary intake was performed at baseline and after two months of intervention. Nutritional assessment was quantitatively and qualitatively performed using a 72 hours' dietary record and food frequency questionnaire (FFQ). Data from food intakes were obtained in the course of individual interviews to request information from each participant about the types of foods and serving sizes. Dietary intake was compared with the daily recommended allowances (DRA). Insufficient intake levels were determined by comparing actual intakes of different nutrients with the recommended intake for each participant and were recorded as below 75% of the RDA. FFQ was used to set the information about the frequency consumption in each group of foods. FFQ was compared with the recommendations proposed by the Spanish Community Nutrition Society (SENC) and expressed as the percentage of participants below or above the recommended servings.
Biochemical parameters - Clinical-nutritional parameters | 2 months
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). The following measurements were taken: Glucose (mg/dL), creatinine (mg/dL), urea (mg/dL), uric acid (mg/dL), triglycerides (mg/dL), total cholesterol (mg/dL), total proteins (g/dL), transferrin (mg/dL) and albumin (mg/dL).
Hormonal parameters | 2 months
  Hormonal parameters were performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®) and determined by colorimetric enzymoimmunoassay techniques (ECLIA, Elecsys 2010 and Modular Analytics E170, Roche Diagnostics, Mannheim, Germany.
  The following measurements were taken: leptin (ng/mL), PTH (pg/mL) and Osteocalcin (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Planells, PhD, Study Director — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vazquez-Lorente H, Molina-Lopez J, Herrera-Quintana L, Gamarra-Morales Y, Quintero-Osso B, Lopez-Gonzalez B, Planells E. Erythrocyte Zn concentration and antioxidant response after supplementation with Zn in a postmenopausal population. A double-blind randomized trial. Exp Gerontol. 2022 Jun 1;162:111766. doi: 10.1016/j.exger.2022.111766. Epub 2022 Mar 9. PMID 35278643